CLINICAL TRIAL: NCT00644969
Title: A Phase 3B 12-Week, Double -Blind, Placebo-Controlled, Multicenter Study Evaluating the Safety and Efficacy of Varenicline Tartrate (CP-526,555) 1 mg BID for Smoking Cessation in Subjects With Schizophrenia and Schizoaffective Disorder.
Brief Title: Smoking Cessation Study for Patients With Schizophrenia or Schizoaffective Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: A3051072
Record Dates: First submitted 2008-03-21; First posted 2008-03-27 (Estimated); Results first posted 2011-04-15 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Arm (Placebo Comparator): Randomization 2:1 treatment to placebo
  Interventions: Drug: placebo
- Treatment Arm (Active Comparator)
  Interventions: Drug: varenicline (CP-526,555)

INTERVENTIONS:
Drug: placebo — Randomization 2:1 treatment to placebo
  Arms: Placebo Arm
Drug: varenicline (CP-526,555) — One week of titration up to 1mg bid and 11 weeks of dosing at 1mg bid
  Other Names: Chantix, Champix
  Arms: Treatment Arm

SUMMARY:
Study will determine whether patients with schizophrenia or schizoaffective disorder can be helped to quit smoking safely while using varenicline and receiving smoking cessation counseling.

DETAILED DESCRIPTION:
This is a safety study.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis (using the SCID-I/P at screening visit) of schizophrenia or schizoaffective disorder and judged to be stable (without hospitalization or acute exacerbation and functioning in society) on psychiatric treatment for at least the past 6 month.
* Current cigarette smokers (at least 15/day during the past year with no period of abstinence greater than 3 months in the past year) male or female, between the ages of 18 and 75 inclusive, who are motivated to stop smoking.
* Score 7 or higher on the Contemplation Ladder at the Screening, Week -1, and Baseline Visits.

Exclusion Criteria:

* PANSS score >70 at Screen or Baseline Visit.
* Subjects hospitalized within the past six months due to suicidal ideation or suicidal behavior or subjects considered to have serious suicidal ideation or suicidal behavior within the past six moth.
* Subjects having active suicidal ideation or behavior identified at Screen, Week -1, or Baseline Visit.
* Subjects taking Bupropion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (9):
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Farmington, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
- Canada (3):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Williams JM, Anthenelli RM, Morris CD, Treadow J, Thompson JR, Yunis C, George TP. A randomized, double-blind, placebo-controlled study evaluating the safety and efficacy of varenicline for smoking cessation in patients with schizophrenia or schizoaffective disorder. J Clin Psychiatry. 2012 May;73(5):654-60. doi: 10.4088/JCP.11m07522. PMID 22697191
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051072&StudyName=Smoking%20Cessation%20Study%20for%20patients%20with%20Schizophrenia%20or%20Schizoaffective%20disorder

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Double-blind treatment phase Week 1 to Week 12. Treatment discontinued at Week 12 and participants continued in Post treatment phase (non-treatment follow up) up to Week 24. Participants could discontinue treatment at any time during treatment phase and remain on study through the non-treatment follow up period.
Groups:
- Varenicline: Varenicline 0.5 milligrams (mg) once a day (QD) for 3 days followed by titration to 0.5 mg twice a day (BID) for 4 days, then 1 mg BID up to Week 12.
- Placebo: Placebo (matching study treatment) 0.5 mg QD for 3 days followed by titration to 0.5 mg BID for 4 days, then 1 mg BID up to Week 12.
Period: Treatment Phase
Arm/Group | Varenicline | Placebo
Started | 85 | 43
Completed | 71 | 40
Not Completed | 14 | 3
Not completed — Randomized, not treated | 1 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 2 | 2
Not completed — Other | 4 | 1
Period: Post Treatment Phase
Arm/Group | Varenicline | Placebo
Started | 71 | 40
Completed | 61 | 37
Not Completed | 10 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 4 | 1
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Placebo | Total
Number analyzed (Participants) | 85 | 43 | 128
Age, Customized [Number; unit: participants]
  18 to 34 years | 33 | 11 | 44
  35 to 44 years | 10 | 9 | 19
  45 to 64 years | 42 | 23 | 65
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 65 | 33 | 98
Number of participants with suicidal behavior and / or ideation on Columbia Suicide Severity Rating [Number; unit: participants] — Clinician rated assessment of suicidal behavior and / or intent: Suicidal behavior=a "yes" response to any of 5 suicidal behavior questions on C-SSRS; Suicidal ideation=a "yes" response to any one of 5 suicidal ideations questions on C-SSRS. Number of participants assessed= 84, 42 for Varenicline and placebo, respectively.
  participants | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AEs are any untoward medical occurrence in a clinical investigation participant administered a product or medical device. The event does not need to be causally related to the study treatment or usage. SAEs include any untoward medical occurrence that results in death, are life threatening, requires hospitalization or prolongation of hospitalization, results in disability or incapacity or are a congenital anomaly or birth defect in the offspring of a study participant. Lack of efficacy was to be reported as an AE when it was associated with an SAE.
Time Frame: Baseline up to 30 days after last dose of study treatment or up to Week 16
Population: Safety analysis set: all participants who took at least 1 dose of randomized study medication, including partial doses and had a safety measurement. Safety assessed Baseline through Week 12 (treatment phase) plus a 30 day lag period after last dose of study treatment).
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
participants
  Serious Adverse Events | 5 | 4
  Adverse Events | 70 | 35

2. Primary Outcome: Number of Participants With Psychiatric Adverse Events
Description: Psychiatric Adverse Event symptoms included, but were not restricted to, depression, anxiety, hostility, perceptual / thinking disturbance, suicidal ideation, or suicidal behavior based on clinical judgment and use of the Positive and Negative Syndrome Scale and Columbia Classification Algorithm of Suicide assessments.
Time Frame: Baseline up to Week 24
Population: Safety analysis set; Safety assessed Baseline through Week 12 (treatment phase) plus a 30 day lag period after last dose of study treatment). Neuropsychiatric events assessed through Week 24.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
participants
  Abnormal dreams | 6 | 4
  Aggression | 0 | 1
  Agitation | 0 | 1
  Anxiety | 4 | 4
  Depressed mood | 2 | 1
  Depression | 4 | 3
  Hallucination auditory | 4 | 1
  Hallucination visual | 1 | 0
  Initial insomnia | 1 | 0
  Insomnia | 8 | 2
  Nervousness | 1 | 0
  Nightmare | 1 | 0
  Panic reaction | 1 | 0
  Paranoia | 2 | 0
  Psychiatric symptom | 1 | 0
  Restlessness | 1 | 0
  Sleep disorder | 1 | 1
  Suicidal ideation | 5 | 3
  Suicide attempt | 1 | 0
  Tension | 1 | 0

3. Primary Outcome: Change From Baseline to Week 12 in Positive and Negative Syndrome Scale (PANSS): Total Score
Description: PANSS includes 30 items rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme) organized as 7 positive symptom subscale items, 7 negative symptom subscale items and 16 general psychopathology items. Total scores range from 30 to 210 with higher scores indicating more extreme symptoms.
Time Frame: Baseline to Week 12
Population: Safety analysis set; (n)=number of participants with analyzable data at observation for varenicline and placebo, respectively.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
scores on a scale
  Baseline mean | 55.88 (9.5) | 54.47 (10.67)
  Mean change at Week 12 (n=68, 39) | -5.19 (8.99) | -3.46 (7.52)

4. Primary Outcome: Change From Baseline to Week 24 in Positive and Negative Syndrome Scale (PANSS): Total Score
Description: as for outcome 3
Time Frame: Baseline to Week 24
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
scores on a scale | -4.77 (10.63) | -3.27 (7.98)

5. Primary Outcome: Change From Baseline to Week 12 in Positive and Negative Syndrome Scale (PANSS): Positive Symptoms Score
Description: PANSS includes 30 items rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme) organized as 7 positive symptom subscale items, 7 negative symptom subscale items and 16 general psychopathology items. Positive symptoms (productive symptoms) associated with schizophrenia (delusions, conceptual disorganization, and hallucinatory behavior) are rated on a scale from 1 (absent) to 7 (extreme); total positive subscale scores range from 7 to 49 with higher scores indicating more extreme symptoms.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
scores on a scale
  Baseline mean | 13.43 (3.23) | 13.53 (4.15)
  Mean change at Week 12 (n=68, 39) | -1.87 (3.34) | -1.33 (2.83)

6. Primary Outcome: Change From Baseline to Week 24 in Positive and Negative Syndrome Scale (PANSS): Positive Symptoms Score
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
scores on a scale | -1.49 (3.8) | -1.68 (2.82)

7. Primary Outcome: Change From Baseline to Week 12 in Positive and Negative Syndrome Scale (PANSS): Negative Symptoms Score
Description: PANSS includes 30 items rated on a 7-point scale (1=absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, 7=extreme) organized as 7 positive symptom subscale items, 7 negative symptom subscale items and 16 general psychopathology items. Negative symptoms (deficit features) associated with schizophrenia (blunted affect, emotional withdrawal, poor rapport, and passive / apathetic social withdrawal) are rated on a scale from 1 (absent) to 7 (extreme); total negative subscale scores range from 7 to 49 with higher scores indicating more extreme symptoms.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
scores on a scale
  Baseline mean | 14.75 (4.12) | 14.79 (4.95)
  Mean change at Week 12 (n=68, 39) | -1 (3.37) | -1.33 (2.97)

8. Primary Outcome: Change From Baseline to Week 24 in Positive and Negative Syndrome Scale (PANSS): Negative Symptoms Score
Description: as for outcome 7
Time Frame: Baseline to Week 24
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
scores on a scale | -1.43 (3.68) | -0.68 (3.76)

9. Primary Outcome: Change From Baseline to Week 12 in Simpson Angus Rating Scale (SARS)
Description: 10-item rating scale to assess the severity of extrapyramidal symptoms rated on a 5-point scale 0 (normal) to 4 (highest severity). Items measured are gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head dropping, glabella tap, tremor, and salivation. Global score calculated by summing individual item scores and dividing by the total number of items; range is 0 to 40 with higher scores indicating greater severity.
Time Frame: Baseline to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
scores on a scale
  Baseline mean | 1.452 (2.061) | 1.139 (1.846)
  Mean change at Week 12 (n=68, 39) | -0.42 (1.341) | 0.102 (1.984)

10. Primary Outcome: Change From Baseline to Week 24 in Simpson Angus Rating Scale (SARS)
Description: as for outcome 9
Time Frame: Baseline to Week 24
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
scores on a scale | -0.37 (1.253) | -0.29 (1.221)

11. Primary Outcome: Number of Participants With Suicidal Behavior and / or Ideation ("Yes" Response) on the Columbia Suicide Severity Rating Scale (C-SSRS) During the Treatment Phase
Description: C-SSRS is a clinician rated assessment of suicidal behavior and / or intent categorized as: Suicidal behavior=a "yes" response to any of 5 suicidal behavior questions (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide); Suicidal ideation=a "yes" response to any one of 5 suicidal ideation questions which includes wish to be dead, and 4 different categories of active suicidal ideation (thought, thought with method, thought with intent, thought with plan and intent).
Time Frame: Week 1 to Week 12 (Treatment phase)
Population: Safety analysis set; N=number of participants assessed for suicidal behavior and / or ideation. "Yes" response includes participants with continued or new suicidal behavior and / or ideation. Treatment phase includes a 7 day lag after last dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 82 | 43
participants | 9 | 4

12. Primary Outcome: Number of Participants With Suicidal Behavior or Suicical Ideation ("Yes" Response ) on the Columbia Suicide-Severity Rating Scale (C-SSRS) During the Post Treatment Phase
Description: as for outcome 11
Time Frame: Week 13 to Week 24 (Post treatment phase)
Population: Safety analysis set; N=number of participants assessed for suicidal behavior and / or ideation. "Yes" response includes participants with new suicidal behavior and / or ideation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 70 | 39
participants | 6 | 0

13. Primary Outcome: Number of Participants With Shift From Baseline to Week 12 in Clinical Global Impressions Scale-Severity (CGI-S) Score
Description: CGI-S: 7-point clinician rated scale to assess severity of participant's current illness state; range: 1=normal, not ill at all, 2=borderline mentally ill, 3=mildly ill, 4=moderately ill, 5=markedly ill, 6=severely ill, 7=among the most extremely ill patients. Higher scores reflect higher severity of current illness states.
Time Frame: Baseline (Bsl) to Week 12
Population: Safety analysis set; N=number of participants with evaluable data at observation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 68 | 39
participants
  Mildly ill Bsl to Borderline ill Week 12 | 1 | 0
  Mildly ill Bsl to Moderately ill Week 12 | 1 | 1
  Moderately ill Bsl to Borderline ill Week 12 | 1 | 0
  Moderately ill Bsl to Mildly ill Week 12 | 4 | 1
  Markedly ill Bsl to Moderately ill Week 12 | 1 | 0

14. Primary Outcome: Number of Participants With Shift From Baseline to Week 24 in Clinical Global Impressions Scale-Severity (CGI-S) Score
Description: as for outcome 13
Time Frame: Baseline to Week 24
Population: Safety analysis set; N=number of participants with evaluable data at observation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
participants
  Mildly ill Bsl to Borderline ill Week 24 | 1 | 0
  Mildly ill Bsl to Moderately ill Week 24 | 1 | 1
  Mildly ill Bsl to Markedly ill Week 24 | 1 | 0
  Moderately ill Bsl to Borderline ill Week 24 | 1 | 0
  Moderately ill Bsl to Mildly ill Week 24 | 5 | 1
  Markedly ill Bsl to Moderately ill Week 24 | 1 | 0

15. Primary Outcome: Number of Participants With Clinical Global Impression of Improvement Scale (CGI-I) Score at Week 1
Description: CGI-I: 7-point clinician rated scale ranging from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, to 7=very much worse. Improvement is defined as a score of 1 (very much improved), 2 (much improved), or 3 (minimally improved) on the scale. Scores above 4 reflect worsening of illness state as compared to baseline.
Time Frame: Baseline, Week 1
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 79 | 43
participants
  Very much improved | 0 | 0
  Much improved | 3 | 0
  Minimally improved | 4 | 3
  No change | 67 | 37
  Minimally worse | 5 | 3
  Much worse | 0 | 0
  Very much worse | 0 | 0

16. Primary Outcome: Number of Participants With Clinical Global Impression of Improvement Scale (CGI-I) Score at Week 12
Description: as for outcome 15
Time Frame: Baseline, Week 12
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 68 | 39
participants
  Very much improved | 1 | 0
  Much improved | 1 | 0
  Minimally improved | 5 | 4
  No change | 55 | 35
  Minimally worse | 6 | 0
  Much worse | 0 | 0
  Very much worse | 0 | 0

17. Primary Outcome: Number of Participants With Clinical Global Impression of Improvement Scale (CGI-I) Score at Week 24
Description: as for outcome 15
Time Frame: Baseline, Week 24
Population: Safety analysis set; N=number of participants with analyzable data at observation.
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 61 | 37
participants
  Very much improved | 2 | 0
  Much improved | 2 | 1
  Minimally improved | 8 | 5
  No change | 46 | 31
  Minimally worse | 2 | 0
  Much worse | 1 | 0
  Very much worse | 0 | 0

18. Secondary Outcome: Number of Participants With 7-day Point Prevalence of Non-smoking at Week 12
Description: 7-day point prevalence of non-smoking measured as the number of participants who maintained complete abstinence from cigarette smoking or other nicotine use in the previous 7 days before the Week 12 visit and had an end-expiratory carbon monoxide (CO) measurement of ≤10 parts per million (ppm).
Time Frame: Week 12
Population: Full analysis set (FAS): all participants randomized into the study who received at least 1 dose of study treatment (formerly referred to as the All subjects analysis set).
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
participants | 16 | 2
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.0457, Regression, Logistic; Odds Ratio (OR) = 4.74, 95% CI 2-sided [1.03 to 21.78]

19. Secondary Outcome: Number of Participants With 7-day Point Prevalence of Non-smoking at Week 24
Description: 7-day point prevalence of non-smoking measured as the number of participants who maintained complete abstinence from cigarette smoking or other nicotine use in the previous 7 days before the Week 24 visit and had an end-expiratory carbon monoxide (CO) measurement of ≤10 parts per million (ppm).
Time Frame: Week 24
Population: FAS
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
participants | 10 | 1
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Test type: Superiority or Other; p = 0.0901, Regression, Logistic; Odds Ratio (OR) = 6.18, 95% CI 2-sided [0.75 to 50.71]

20. Secondary Outcome: Number of Participants With at Least a 50 Percent (%) Reduction From Baseline to Week 12 and Week 24 in the Number of Cigarettes Smoked Per Day
Description: Measured as at least a 50% reduction from baseline in cigarettes smoked per day averaged over the past 7 days at Week 12 and Week 24.
Time Frame: Baseline, Week 12, Week 24
Population: FAS
Measure: Number; unit: participants
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
participants
  Week 12 | 54 | 22
  Week 24 | 34 | 18
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12; Test type: Superiority or Other; p = 0.1524, Regression, Logistic; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.82 to 3.68]
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24; Test type: Superiority or Other; p = 0.9235, Regression, Logistic; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.45 to 2.05]

21. Secondary Outcome: Change From Baseline to Week 12 and Week 24 in the Number of Cigarettes Smoked Per Day
Description: Measured as mean number of cigarettes smoked per day averaged over the past 7 days at Week 12 and Week 24.
Time Frame: Baseline, Week 12, Week 24
Population: FAS; (n)=number of participants with evaluable data at observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: cigarettes per day
Arm/Group | Varenicline | Placebo
Number analyzed (Participants) | 84 | 43
cigarettes per day
  Week 12 (n=68, 39) | -14.23 [-15.95 to -12.51] | -10.58 [-12.73 to -8.42]
  Week 24 (n=61, 37) | -9.55 [-12.00 to -7.10] | -9.32 [-12.36 to -6.28]
Statistical Analysis 1: Comparison: Varenicline vs Placebo; Week 12 treatment difference; Test type: Superiority or Other; p = 0.0077, ANCOVA; Mean Difference (Final Values) = -3.65, 95% CI 2-sided [-6.32 to -0.99] — Least squares mean difference
Statistical Analysis 2: Comparison: Varenicline vs Placebo; Week 24 treatment difference; Test type: Superiority or Other; p = 0.9022, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-3.99 to 3.52] — Least squares mean difference

ADVERSE EVENTS:
Time Frame: Events assessed Baseline through Week 12 (treatment phase) plus a 30 day lag period after last dose of study treatment); Neuropsychiatric events assessed through Week 24.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline | Placebo
Serious Adverse Events (participants affected / at risk) | 5/84 | 4/43
Other Adverse Events (participants affected / at risk) | 48/84 | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=84) | Placebo (N=43)
Chest pain (General disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Aggression (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Psychiatric symptom (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=84) | Placebo (N=43)
Abdominal pain upper (Gastrointestinal disorders) | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 20 | 6
Vomiting (Gastrointestinal disorders) | 9 | 4
Fatigue (General disorders) | 5 | 2
Irritability (General disorders) | 5 | 3
Upper respiratory tract infection (Infections and infestations) | 6 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Headache (Nervous system disorders) | 9 | 8
Abnormal dreams (Psychiatric disorders) | 6 | 4
Anxiety (Psychiatric disorders) | 4 | 4
Depression (Psychiatric disorders) | 3 | 3
Insomnia (Psychiatric disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.